CLINICAL TRIAL: NCT03576937
Title: Achieving Value in Cancer Diagnostics: Blood Versus Tissue Molecular Profiling - a Prospective Canadian Study
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5353
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with advanced (incurable stage IIIB or IV), histologically proven, non-squamous NSCLC who are never- or light-smokers (≤10 pack year smoking history) and are being considered for systemic therapy in the first line setting are eligible. Blood will be collected prior to first line treatment for testing cfDNA with the GUARDANT360 assay. Testing of available diagnostic tissue for genomic abnormalities will be performed in all patients per standard of care at the participating sites.
  Interventions: Diagnostic Test: GUARDANT360
- Cohort 2: Patients with advanced non-squamous NSCLC with known oncogenic drivers (such as EGFR, ALK, ROS-1, BRAF) that have failed tyrosine kinase inhibitor (TKI) therapy, and are being considered for subsequent therapy. Blood will be collected from patients at time of progression on TKI therapy for cfDNA testing with the GUARDANT360 assay. Testing of available diagnostic tissue for genomic abnormalities will be performed in all patients per standard of care at the participating sites.
  Interventions: Diagnostic Test: GUARDANT360

INTERVENTIONS:
Diagnostic Test: GUARDANT360 — GUARDANT360 is a validated cfDNA next-generation sequencing assay that identifies variants in 73 genes associated with several cancers.

SUMMARY:
Current guidelines in non-small cell lung cancer recommend genomic assessment for mutations in EGFR and BRAF, gene rearrangements in ALK and ROS1, and resistance mutations such as T790M upon progression during EGFR inhibitor therapy. However, obtaining sufficient tumour tissue to test for these molecular alterations, as well as those with emerging targeted therapies, is challenging in lung cancer. A promising method to improve molecular diagnostic testing in lung and other cancers is the use of circulating cell-free DNA (cfDNA) obtained from blood samples or liquid biopsies. This multi-centre prospective study will compare blood-based profiling (using the GUARDANT360 assay) to standard of care tissue-based profiling within the Canadian system.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-small cell lung cancer (NSCLC) with:

1. Histologically-proven, advanced (Stage IIIB or IV not eligible for curative intent treatment, or relapsed/recurrent) disease;
2. Non-squamous histology (mixed adenocarcinoma histology is allowed);
3. Never smoking or light smoking history (≤10 pack years);
4. Measureable disease by RECIST 1.1;
5. Patients who have previously received curative therapy are eligible if primary treatment was completed at least 6 months prior to the development of advanced disease; for patients who received adjuvant systemic therapy, the last dose of treatment must have been given at least 6 weeks prior to enrollment;
6. Age ≥ 18 years;
7. Ability to provide written informed consent;
8. Agreement to provide blood sample prior to starting systemic treatment;
9. Eligibility for targeted therapy in the opinion of the investigator;
10. Standard-of-care tissue genotyping ordered or planned. Patients with tissue deemed insufficient for genotyping are eligible.
11. Cohort 2 only: evidence of disease progression on prior targeted tyrosine kinase inhibitor or other targeted therapy for EGFR including T790M, ALK, ROS-1 or BRAF-deranged advanced NSCLC. Patients progressing on 1st or 2nd generation EGFR TKI must have undergone SOC testing for EGFR T790M. If blood- or tissue-negative for T790M, the patient is eligible for this study. If T790M-positive, the patient must have progressed on a T790M inhibitor to be eligible. Intervening systemic therapy such as chemotherapy or immunotherapy is permitted.

Exclusion Criteria:

1. Pregnancy;
2. ≥10 pack year smoking history;
3. Any other concurrent malignancy except for localized, non-melanoma, cutaneous cancer or non-invasive cervical cancer. Any prior cancer other than NSCLC must have occurred more than 2 years prior to study entry with no evidence of currently active disease;
4. Prior resection of metastatic disease if the resected metastasis was the only site of measurable disease;
5. Radiation of a metastatic lesion or residual disease if administered to the only site(s) of advanced disease;
6. Cohort 1 only: Prior systemic treatment for metastatic NSCLC including but not limited to targeted therapy, chemotherapy, immunotherapy, or biologic therapy. Adjuvant therapy is permitted at least 6 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients (Stage IIIB or IV not eligible for curative intent treatment, or relapsed/recurrent disease)
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Response rate to first-line therapy | Up to 18 Months
  Measure best response to first-line therapy using investigator-assessed RECIST 1.1, including progression free survival and time to treatment failure, in patients with advanced lung adenocarcinoma using the cfDNA GUARDANT360 assay versus standard of care tissue genotyping.

SECONDARY OUTCOMES:
Proportion of patients receiving targeted therapy | Up to 18 Months
  Compare the proportion of patients receiving targeted therapy using the cfDNA GUARDANT360 assay versus standard of care tissue genotyping.
Time to Treatment Initiation | Up to 18 Months
  The time to treatment initiation using both genotyping methods, will be calculated as the number of days from the date of pathologic or clinical stage IV NSCLC diagnosis until initiation of systemic treatment. This will be compared to the turnaround time for GUARDANT360 results.
Incremental number of actionable genomic alterations | Up to 18 Months
  Count the number of actionable genomic alterations identified in cfDNA that were not identified in tumour tissue standard of care testing.
Turnaround time of cfDNA vs. tissue results | Up to 18 Months
  Calculate the time (in days) from the date of request for testing to the report date for both genotyping methods.
Costs of cfDNA vs. tissue testing | Up to 18 Months
  Cost consequence analysis to examine incremental mean direct and indirect costs in Canadian dollars between the two approaches (cfDNA testing vs tumour tissue genotyping).

OTHER OUTCOMES:
Response rate to immunotherapy | Up to 18 Months
  Assess response rate in patients (Cohort 1) who received single agent or combination immunotherapy.
Response duration to immunotherapy | Up to 18 Months
  Assess response duration in patients (Cohort 1) who received single agent or combination immunotherapy.
Patient reported quality of life | Upon entry and 3 months following initiation of systemic therapy
  Patient quality of life will be measured using the EQ5D-5L, which will be administered upon entry to the study and 3 months after starting systemic therapy.
Patient willingness-to-pay | Within 30 days of study enrollment
  Evaluate patient willingness-to-pay for using a next generation sequencing assay, such as the GUARDANT360, using a validated patient survey.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No